CLINICAL TRIAL: NCT07366515
Title: Feasibility of a Multimodal Virtual Reality Intervention to Reduce Preoperative Anxiety in Cancer Surgery Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Renée El-Gabalawy, Associate Professor & Clinical Psychologist, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 0414
Record Dates: First submitted 2025-12-10; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Oncologic Surgery
Keywords: virtual reality; oncological surgery; feasibility; perioperative mental health; preoperative anxiety and distress

STUDY DESIGN:
Intervention Model Description: All participants will engage in a single in-person virtual reality session approximately two weeks prior to their surgery. After the session, all participants will be provided with a link to a standardized recorded virtual reality session allowing them to review the intervention experience. Half of the participants will be instructed to watch the video daily, while the other half will be instructed to watch the video at their discretion.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily Viewing Group (Other): Participants assigned to this group will be instructed to review the standardized VR intervention recording daily, following their in-person session and continuing up to their scheduled surgery date.
  Interventions: Device: Virtual Reality
- Self-directed group (Other): Participants assigned to this group will be instructed to review the standardized VR intervention recording as little or as much as they would like, following their in-person session and continuing up to their scheduled surgery date.
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — The VR simulation involves the experience of prepping, waiting, receiving, and recovering from surgery at a large tertiary care centre in Central Canada. It is designed to prepare patients for cancer surgery by increasing familiarity with the hospital environment, providing the opportunity to "experience" restricted areas of the hospital that patients cannot access until the day of the surgery, and better understand the surgical process. The simulation was originally developed for a prior research project focused on breast cancer surgery and has since been adapted based on participant feedback. The intervention includes multiple modules that progress from an orientation to the hospital environment to more immersive, first-person surgical experiences.

SUMMARY:
The goal of this study is to assess the feasibility of an expanded virtual reality (VR) intervention designed to help prepare patients for cancer surgery. This study will: (1) assess the investigator's ability to recruit, retain, and engage participants, (2) evaluate how acceptable participants find the intervention through their feedback on its individual components. The investigators will also explore whether baseline anxiety levels or psychiatric history predict responses to the intervention, as well as look for any changes in perioperative anxiety and monitoring for any adverse effects associated with the intervention. This study will also investigate engagement of providing participants with a first-person VR session recordings to determine utility and whether post-session access is perceived as beneficial. Finally, preliminary pilot outcomes will examine whether increased engagement in the VR results in reductions in anxiety on the day of surgery.

ELIGIBILITY:
Patients will be deemed eligible for inclusion if they: (a) are 18 years of age or older; (b) are able to speak and read English; (c) have received a cancer diagnosis; and (d) are scheduled, or in the process of being scheduled to undergo oncological surgery under general anesthesia at the Health Sciences Centre Winnipeg. Patients will be deemed ineligible if they are unable to provide informed consent (e.g., due to cognitive impairment) or if they have any visual, auditory and/or motor impairments that would preclude effective participation in the Virtual Reality intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Engagement | Day 0 post-intervention
  Length of time in minutes participants spent engaging with the virtual reality and each of its components during the in-person session
Acceptability | Day 0 post-intervention
  The Theoretical Framework of Acceptability Questionnaire (TFAQ score > 3 indicates acceptability). Range 1-5 on seven items.

SECONDARY OUTCOMES:
Anxiety | Baseline
  Generalized Anxiety Disorder 7. Range 0 to 21, higher score = higher anxiety.
Depression | Baseline
  Patient Health Questionnaire-8 (PHQ-8). Range 0 to 24, higher score = higher depressive symptoms.
Pre-Operative Anxiety | Baseline and re-administered pre-operatively on the day of surgery
  Amsterdam Preoperative Anxiety and Information Scale (APAIS). Range 4 - 30 for 6 items.
Pre-Operative Anxiety | Baseline
  Pre-operative Intrusive Thoughts Inventory (PITI). Range 0 to 60 on 20 items, score >15 indicative of clinically significant preoperative anxiety.
Pre-Operative Anxiety | Baseline and re-administered pre-operatively on the day of surgery.
  National Comprehensive Cancer Network (NCCN) Anxiety Thermometer. A brief self-report visual analogue scale (VAS) for anxiety. Range 0 to 10, higher score = higher anxiety
Pre-Operative Distress | Baseline and re-administered pre-operatively on the day of surgery
  NCCN Distress Thermometer. A brief self-report visual analogue scale (VAS) for anxiety. Range 0 to 10, higher score = higher distress.
Cybersickness | Day 0 post-intervention
  Simulator Sickness Questionnaire. Range 0-3 for each 16 items, higher score = more severe symptoms.
Presence | Day 0 post-intervention
  iGroup Presence Questionnaire. Range -3 to +3 for each of 14 items, higher score = higher presence.
Perceived Usability of Device | Day 0 post-intervention
  System Usability Scale. Range 1 to 5 for each of 10 items, higher score = better usability
Engagement & Adherence - Standardized Video | Day 1 up to Day 14
  Length of time in minutes that the participant engaged with the standardized video, and whether this aligned with the instructions provided.

CONTACTS AND LOCATIONS:
Overall Officials: Renee El-Gabalawy, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared, consistent with common practice in feasibility studies.